CLINICAL TRIAL: NCT06606626
Title: Relationship Between Sleep Time and Quality With the Production of Force, Power, and Muscular Endurance.
Brief Title: Sleep and Resistance Exercise
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alcala (Other)
Responsible Party: Principal Investigator, Alberto Pérez-López, Principal Investigator, University of Alcala
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Other
Other Study IDs: CEID/2023/6/119
Record Dates: First submitted 2024-09-09; First posted 2024-09-23 (Actual); Last update posted 2025-05-25 (Actual); Status verified 2025-05

CONDITIONS: Sleep Deprivation
MeSH Terms: conditions — Sleep Deprivation

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: Statistician
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- 8h Sleep (at home) (Placebo Comparator): Participants sleep 8h at home
  Interventions: Behavioral: Sleep place
- 8h Sleep (Laboratory) (Experimental): Participants sleep 8h in the lab
  Interventions: Behavioral: Sleep deprivation; Behavioral: Sleep place
- 4h Sleep (Laboratory) (Experimental): Participants sleep 4h in the laboratory
  Interventions: Behavioral: Sleep deprivation
- 0h Sleep (Laboratory) (Experimental): Participants sleep 0h in the laboratory
  Interventions: Behavioral: Sleep deprivation

INTERVENTIONS:
Behavioral: Sleep deprivation — Partial (4h) or total (0h) sleep deprivation
  Arms: 0h Sleep (Laboratory); 4h Sleep (Laboratory); 8h Sleep (Laboratory)
Behavioral: Sleep place — 8h sleep at home or in the laboratory
  Arms: 8h Sleep (Laboratory); 8h Sleep (at home)

SUMMARY:
Introduction: Despite the awareness of the importance of sleep in our lives, especially for athletes, the consequences of poor rest on sports performance are not well understood. Furthermore, the interaction between complete and partial sleep deprivation over one night and sleeping the usual hours for each person remains unclear.

Objectives: The aim of this study is to evaluate the effects of sleep deprivation on the production of strength, power, and muscular endurance according to sex (men vs. women) and type of exercise (bench press vs. squat). Additionally, the study will analyze the effects of sleep deprivation on perceived fatigue, mood, dietary habits, electrical activity, resting metabolic rate (RMR), and maximal fat oxidation (MFO).

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 35 years.
* Body Mass Index (BMI) < 25 kg/m².
* Resistance-trained individuals (more than 2 years of structured training).
* Healthy men and women without neurological, cardiometabolic, immunological, or physical conditions that prevent them from exercising.
* Participants must be able to perform the tests described in the following section.

Exclusion Criteria:

* History of neuromuscular diseases, heart disease, or conditions that may affect liver or muscle metabolism.
* Use of drugs, stimulants, or sports supplements that could interfere with the dietary supplement used in the study.
* Sedentary habits (less than 150 minutes/week of moderate exercise).
* Having undergone prolonged periods of physical inactivity in the 6 months prior to the study.
* Engaging in strenuous exercise within 48 hours prior to the tests.
* Failure to replicate the same food intake on both experimental days.
* Consumption of caffeine or any other stimulant the day before the tests.

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 28 (Actual)
Dates: Start 2024-01-07 (Actual); Primary Completion 2025-01-30 (Actual); Study Completion 2025-01-30 (Actual)

PRIMARY OUTCOMES:
Mean velocity at different %1RM | Through study completion, an average of 4 weeks
  Measuring bar mean velocity desplacement during bench press and back squat exercises.
Peak velocity at different %1RM | Through study completion, an average of 4 weeks
  Measuring bar peak velocity and time to reach peak velocity of bar desplacement during bench press and back squat exercises.
Mean power output at different %1RM | Through study completion, an average of 4 weeks
  Measuring during bench press and back squat exercises.
Peak power output and time to reach peak power output at different %1RM | Through study completion, an average of 4 weeks
  Measuring during bench press and back squat exercises.
Number of repetitions performed at 65%1RM until task failure | Through study completion, an average of 4 weeks
  In bench press and back squat exercises
Bar velocity deplacement performed in 1 set at 65%1RM until task failure | Through study completion, an average of 4 weeks
  In bench press and back squat exercises
Power output generated in 1 set at 65%1RM until task failure | Through study completion, an average of 4 weeks
  In bench press and back squat exercise
Resting Metabolic Rate (RMR) | Through study completion, an average of 4 weeks
  Kcal at rest measuring a metabolic chart
Maximal Fat Oxidation Rate | Through study completion, an average of 4 weeks
  g/min using a metabolic chart

SECONDARY OUTCOMES:
Physical activity (METs-min/wk) | Before each trial, during the 4 weeks
  Using IPAQ
Dietary habits (g/kg of macronutrients) | Before each trial, during the 4 weeks
  Using a 24-total recall
Fat mass | Through study completion, an average of 4 weeks
  Using electrical bioimpedance (kg and % of body mass)
Fat-free mass | Through study completion, an average of 4 weeks
  Using electrical bioimpedance (kg and % of body mass)
Mood state (tension, depression, anger, vigor, fatigue and confusion) | Through study completion, an average of 4 weeks
  Participants graded a set of 29 items related to the mood on a Likert scale from 0 (not at all) to 4 (extremely) in reply to the question;How do you feel at this moment?; to assess six scales: tension, depression, anger, vigor, fatigue and confusion.

CONTACTS AND LOCATIONS:
Locations (1):
- Facultad de Medicina y Ciencias de la Salud. Universidad de Alcalá, Alcalá de Henares, Madrid, Spain

IPD SHARING:
Plan to Share IPD: Yes